CLINICAL TRIAL: NCT06274463
Title: Effects of Customized Trunk Stabilization Exercise Program to Patients With Brain Disease on Trunk Stability and Satisfaction With the Program
Brief Title: A Personalized Trunk Stability Exercise Program Study With Brain Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11-035
Record Dates: First submitted 2024-02-04; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Brain Diseases
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain disease (Experimental)
  Interventions: Behavioral: Exercise therapy including a trunk stabilization exercise program

INTERVENTIONS:
Behavioral: Exercise therapy including a trunk stabilization exercise program — All patients will undergo 30 sessions of exercise therapy, including a trunk stability exercise program, for 30 minutes per day, 5 days a week for 6 weeks

SUMMARY:
To investigate the effect on improving trunk stability and satisfaction with the program when a customized trunk stabilization exercise program personalized to the subject's functional level is applied to patients with brain disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years old
2. Brain disease patients hospitalized in the rehabilitation medicine department of our hospital and receiving exercise therapy 5 times a week
3. Patients with a functional ambulatory category (FAC) score of 0-4
4. After receiving a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to follow the precautions.

Exclusion Criteria:

1. Those who have suffered prior to participating in the study
2. Those in good physical condition, such as unstable conditions in the state system, coordination system, problem system, and endocrine system, and those with cerebrovascular disease
3. Other cases of investigation without participation in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-21 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale | baseline, 5 weeks after intervention
  Trunk impairment scale assessment for motor function of upper extremity in score.
  This evaluation consists of a total score of 23 points and consists of static sitting balance, dynamic sitting balance, and co-ordination. The higher the score, the better the upper extremity motor function.
Berg Balance Scale | baseline, 5 weeks after intervention
  Berg balance scale assessment of balance function by score. It consists of a total of 14 items and is divided into three parts: sitting, standing, and posture change. The minimum score is 0 points, up to 4 points for discharge, and the total total score is 56 points. A higher score means higher balance ability and lower risk of falling.

SECONDARY OUTCOMES:
Joint angle | baseline, 5 weeks after intervention
  Motion analysis is a process of measuring and evaluating kinematic parameters of joint angle(degree) of each joint through Qualisys motion analysis system.
Joint moment | baseline, 5 weeks after intervention
  Evaluating kinetic parameters of joint moment (Nm/kg) of each joint through Qualisys motion analysis system.
Joint power | baseline, 5 weeks after intervention
  Evaluating kinetic parameters of joint power(Nm/s*Kg) of each joint through Qualisys motion analysis system.

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, MD, PhD, Principal Investigator — CHA Bundang Medical Center